CLINICAL TRIAL: NCT07204756
Title: HOPE-BP 2.0: Evaluating the Optimal Duration of Postpartum Remote Blood Pressure Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OBGYN-2025-34107
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postpartum; Hypertension; Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Hypertension; Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-Week Arm (Active Comparator): Participants randomized into the 2 week arm will be immediately unenrolled from the postpartum remote blood pressure monitoring program and resume standard postpartum care
  Interventions: Diagnostic Test: 2-Week Home Monitoring
- 6-Week Arm (Active Comparator): Patients randomized into the 6 week arm will continue and complete the program in its entirety per current SOC (4 additional weeks)
  Interventions: Diagnostic Test: 6-Week Home Monitoring

INTERVENTIONS:
Diagnostic Test: 2-Week Home Monitoring — Those who are randomized into the 2-week intervention arm will be unenrolled from the postpartum remote blood pressure monitoring program and therefore will no longer be transmitting twice daily blood pressures for review.
  Arms: 2-Week Arm
Diagnostic Test: 6-Week Home Monitoring — HOPE-BP provides remote monitoring for the 35% of approximately 2,800 annual births at our institution complicated by HDP. Eligible patients enroll at hospital discharge into a 6-week program, submitting blood pressure readings twice daily via Epic's MyChart Care Companion. Participants receive immediate automated feedback, and a dedicated Maternal Fetal Medicine nursing team reviews data daily (Monday-Friday, 8 AM-4 PM), initiating or adjusting antihypertensive therapy as needed.
  Arms: 6-Week Arm

SUMMARY:
Postpartum remote blood pressure monitoring programs for patients with hypertensive disorders of pregnancy (HDP) are becoming part of standard postpartum management. Existing programs range in duration from 2 to 6 weeks but there has not been any evaluation as to what program duration is optimal. The primary objective of this study is to evaluate the impact of program duration on clinical outcomes for patients participating in a single institution's postpartum remote blood pressure monitoring program for patients with HDP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Discharged after delivery at University of Minnesota Medical Center
* Enrolled into the HOPE-BP Program

Exclusion Criteria:

* Ongoing antihypertensive medication use at 2 weeks (time of randomization)
* Have a medical comorbidity that would not be clinically appropriate to randomize
* Patients opted out of clinical research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Diastolic Blood Pressure | Week 6
  The primary outcome will be the patient's diastolic blood pressure (DBP) at their 6-week postpartum visit.

SECONDARY OUTCOMES:
Systolic Blood Pressure at 6 weeks post-partum | Week 6
  Patient's systolic blood pressure at their 6-week postpartum visit
6-Week Post-partum Follow-up Rates | Week 6
  Participants who complete a 6-week post-partum visit / Total participants eligible for a 6-week post-partum visit
Unscheduled OB visit, triage visit, ED visit, or readmission rates | Week 6
Patient Satisfaction Survey responses at 6 weeks | Week 6
  PSS Score, where higher score indicates greater satisfaction
Rate of severe hypertension | Week 6
  defined as systolic blood pressure ≥ 160mmHg and/or DBP ≥ 110 mmHg
Rate of new hypertension diagnosis at 6 weeks postpartum | Week 6
  based on American Heart Association and American College of Cardiology criteria (AHA/ACC)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Sabol, MD MAS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No